CLINICAL TRIAL: NCT03151083
Title: Implementing and Evaluating Computer-Based Interventions for Mental Health (CDA 14-420)
Brief Title: Implementing and Evaluating Computer-Based Interventions for Mental Health: Testing an Implementation Strategy for VA Outpatient Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 16-001
Record Dates: First submitted 2017-04-19; First posted 2017-05-12 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Insomnia
Keywords: Health Technology; Internet-Based Psychotherapy; self-care; Primary Care; Mental Health
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will employ a hybrid type 3 implementation-effectiveness study design through which the investigator will primarily test the effectiveness of the experimental implementation strategy the investigators are developing and secondarily evaluate the clinical effectiveness of the internet-based self-help program for insomnia. The investigators will use a quasi-experimental pre-/post-cohort design whereby the program will initially be implemented using an enhanced usual care (control) strategy, followed by implementation using the experimental implementation strategy. The program's association with clinical response will be evaluated in an uncontrolled pre-/post-format.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1: Implementation As Usual (Implementation Through Rese (Active Comparator): SHUTi digital CBTi Program was implemented in VACT primary care using implementation activities executed by the research team between June 2017 and January 2018 (8-months). Implementation activities included: Provider Education by the research team, Provider Reminders (information pamphlets in treatment rooms), Patient Advertising/Information (information pamphlets in treatment rooms), Single Referral Pathway Not Integrated Primary Care Workflow (Primary care provider contact research team for patient referral over email).
  Interventions: Behavioral: Internet-based Self-help Insomnia Intervention
- Phase 2: Primary Care Coached Digital CBTi Implementation (Im (Experimental): SHUTi digital CBTi Program implemented in VACT primary care using implementation activities executed by primary care teams June 2018 and January 2019 (8-months). Implementation activities included: Provider Education by the research team, Provider Reminders (information pamphlets in treatment rooms), Patient Advertising/Information (information pamphlets in treatment rooms), patient education and motivational support supplied through a digital CBTi coach, the digital CBTi coach was a primary care nurse trained by the research team, technical support and oversight of the digital CBTi coach by the research team. Single Referral Pathway Not Integrated Primary Care Workflow.
  Interventions: Behavioral: Internet-based Self-help Insomnia Intervention
- Phase 3: Primary Care Mental Health Collaborative Care Implem (Experimental): SHUTi digital CBTi Program implemented in VACT primary care using implementation activities executed by primary care teams April 2019 and November 2019 (8-months). Implementation activities included: Provider Education by the research team, Provider Reminders, Patient Advertising/Information, patient education and motivational support supplied through a digital CBTi coach, the digital CBTi coach was a peer support specialist working on the primary care mental health collaborative care team, the digital CBTi coach was trained by the research team, technical support and oversight of the digital CBTi coach by the research team. Additional members primary care mental health collaborative care team were educated to provide education about digital CBTi. Multiple referral pathways to digital CBTi: consults to the digital CBTi Coach, warm handoffs to primary care mental health collaborative care team. Digital CBTi coach consults integrated Primary Care Workflow.
  Interventions: Behavioral: Internet-based Self-help Insomnia Intervention

INTERVENTIONS:
Behavioral: Internet-based Self-help Insomnia Intervention — The investigators will use the program, SHUTiTM for the treatment of insomnia. The intervention is a CBT-based 6-week, self-administered course accessed via the Internet on mobile, desk-top, and other devices. The program is split into six modules, completed weekly, which include instruction on psycho-education, stimulus control, relaxation training, sleep restriction, medication tapering, and addressing cognitive distortions. The content is delivered via text, video vignettes, case histories, interactive learning tools, interactive skills assessments, symptom assessments, and a sleep log. Homework is assigned after each module. Providers and support staff can follow treatment progress via access to a dashboard of patient information collected by the program. Such information includes progress through the modules, date of last engagement, symptom assessment outcomes, and sleep log data abstracted into commonly used sleep indices such as sleep onset latency and sleep efficiency.
  Other Names: SHUTi (Sleep Health Using the Internet)

SUMMARY:
Internet-based self-help programs are personalized, self-guided interventions delivered over a computer, mobile device, or other Internet platform and focused on improving knowledge, awareness, or behavior change for a mental or physical health problem. Through previous and on-going projects at VACT, the investigators are developing a general strategy for implementing Internet-based Self-help programs in VA primary care, specifically among Patient Aligned Care Teams (PACT) and Primary Care Mental Health Integration (PCMHI) providers. An implementation strategy is defined as a systematic intervention to integrate evidence-based health innovations into usual care. The strategy the investigators propose to test consists of four core components: (1) a clinical intermediary for patient support, (2) provider/staff facilitation and education, (3) patient education, and (4) stepped-care for those requiring additional treatment. In the proposed study, the investigators will compare this strategy to a low intensity (control) strategy with respect to the implementation related outcomes of patent engagement, provider adoption through referral to the program, and patient completion, over a six-month active implementation period. The investigators will target the very common clinical problem of insomnia and use the SHUTiTM program, a 6-week self-guided program utilizing standard cognitive-behavioral therapy (CBT) techniques for the treatment of chronic insomnia. The program has been shown to improve insomnia severity and other sleep related outcomes in a number of controlled trials. The clinical effectiveness of SHUTiTM will be evaluated using clinical insomnia outcomes obtained on all patients enrolled over the 6-month active implementation periods. The purpose this study is to evaluate the preliminary (1) effectiveness of an implementation strategy for Internet-based Self-help Interventions and (2) clinical outcomes of a specific Internet-based self-help program for insomnia, SHUTiTM, in VA Connecticut outpatient primary care. The primary hypothesis is that the experimental implementation strategy the investigators are developing, relative to a control strategy, will result in higher rates of program engagement by patients, greater provider adoption through referral to the program, greater program completion, and improved patient insomnia outcomes.

DETAILED DESCRIPTION:
Objective: The purpose this study is to evaluate the preliminary (1) effectiveness of an implementation strategy for Internet-based Self-help Interventions and (2) clinical outcomes of a specific Internet-based self-help program for insomnia, SHUTiTM, in VA Connecticut outpatient primary care. The primary hypothesis is that the experimental implementation strategy the investigators are developing, relative to a control strategy, will result in higher rates of program engagement by patients, greater provider adoption through referral to the program, greater program completion, and improved patient insomnia outcomes.

Research Design: The investigators will employ a hybrid implementation-effectiveness study design through which the investigators will primarily test the effectiveness of the implementation strategy, while secondarily evaluating the clinical effectiveness of the SHUTiTM program. The investigators will use a quasi-experimental pre-/post-cohort design whereby SHUTiTM will initially be implemented using a low-intensity (control) strategy, followed by implementation using the experimental strategy. The SHUTiTM program's association with clinical response will be evaluated in an uncontrolled pre-/post-format.

Methodology: Internet-based self-help programs are personalized, self-guided interventions delivered over a computer, mobile device, or other Internet platform and focused on improving knowledge, awareness, or behavior change for a mental or physical health problem. Through previous and on-going projects at VACT, the investigators are developing a general strategy for implementing Internet-based Self-help programs in VA primary care, specifically among Patient Aligned Care Teams (PACT) and Primary Care Mental Health Integration (PCMHI) providers. An implementation strategy is defined as a systematic intervention to integrate evidence-based health innovations into usual care. The strategy the investigators propose to test consists of four core components: (1) a clinical intermediary for patient support, (2) provider/staff facilitation and education, (3) patient education, and (4) stepped-care for those requiring additional treatment. The investigators' currently approved protocol (#0002) involves interviewing VA providers, administrators, and staff in order to expand and modify the components of this strategy. In the proposed study, the investigators will compare this strategy to a low intensity (control) strategy with respect to the implementation related outcomes of patent engagement, provider adoption through referral to the program, and patient completion, over a six-month active implementation period. Use of the program will continue and implementation outcomes will be gathered over an additional one-year sustainment phase. The investigators will target the very common clinical problem of insomnia and use the SHUTiTM program, a 6-week self-guided program utilizing standard cognitive-behavioral therapy (CBT) techniques for the treatment of chronic insomnia. The program has been shown to improve insomnia severity and other sleep related outcomes in a number of controlled trials. The clinical effectiveness of SHUTiTM will be evaluated using clinical insomnia outcomes obtained on all patients enrolled over the 6-month active implementation periods.

Impact/Significance: The development and testing of evidence-based implementation strategies for Internet-based self-help programs in VA outpatient care is essential given that (1) there is an increasing number of Internet-based self-help programs providing evidence-based treatment for a variety of mental and behavioral health disorders, (2) VA has committed to improving access to care, especially evidence-based and self-care resources, and (3) there is a Congressional mandate that VA implement Internet-based care. This will be first controlled trial of an implementation strategy for Internet-based self-help programs in a VA primary care (PACT/PCMHI) context.

ELIGIBILITY:
Inclusion Criteria:

* Patients Receiving care from a VA Connecticut West Haven PACT/PCMHI Provider
* Diagnosed with insomnia lasting 3 months by the PACT provider, as evidenced by referral by the provider for access to the SHUTiTM program
* Able to provide valid informed consent, as evidenced by answering questions indicating their understanding of the content of the Informed Consent Document
* Willing to participate in an internet-based self-help program for insomnia after the access to and requirements of the program are explained to them
* English-speaking (The SHUTiTM program is only available in English)

Exclusion Criteria:

* Evidence of acute psychiatric decompensation requiring inpatient admission or emergency department services within the last month, including suicidality, homicidally, mania, or psychotic decompensation.
* Evidence of a conservator of person either verbally reported by the patient or upon inspection of the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hermes, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hermes EDA, Rosenheck RA, Burrone L, Dante G, Lukens C, Martino S. The Implementation and Effectiveness of Digital Cognitive Behavioral Therapy for Insomnia in Primary Care: A Pilot Study. Implement Res Pract. 2021 Nov 15;2:26334895211053659. doi: 10.1177/26334895211053659. eCollection 2021 Jan-Dec. PMID 37090002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment to digital CBTi occurred through primary care providers who made a referrals to the intervention. Referrals were addressed by the digital intervention coach (or research team member, depending on the cohort), who provided and initial education session about digital CBTi. Participants could then enroll in the trial if they wished. Over the entire course of the trial, 153 individuals were referred and 77 chose to enroll.
Groups:
- Phase 1: Implementation As Usual (Implementation Through Research Team): SHUTi digital CBTi Program was implemented in VACT primary care using implementation activities executed by the research team (June 2017 - January 2018). Implementation activities included: Provider Education by the research team, Provider Reminders (information pamphlets in treatment rooms), Patient Advertising/Information (information pamphlets in treatment rooms), Single Referral Pathway Not Integrated Primary Care Workflow (Primary care provider contact research team for patient referral over email).
- Phase 2: Primary Care Coached Digital CBTi Implementation (Implementation Through Primary Care): SHUTi digital CBTi Program implemented in VACT primary care using implementation activities executed by primary care teams (June 2018 to January 2018). Implementation activities included: Provider Education by the research team, Provider Reminders (information pamphlets in treatment rooms), Patient Advertising/Information (information pamphlets in treatment rooms), patient education and motivational support supplied through a digital CBTi coach, the digital CBTi coach was a primary care nurse trained by the research team, technical support and oversight of the digital CBTi coach by the research team. Single Referral Pathway Not Integrated Primary Care Workflow (Primary care provider contact research team for patient referral over email).
- Phase 3: Primary Care Mental Health Collaborative Care Implementation: SHUTi digital CBTi Program implemented in VACT primary care using implementation activities executed by primary care teams (April 2019 to November 2019). Implementation activities included: Provider Education by the research team, Provider Reminders (information pamphlets in treatment rooms), Patient Advertising/Information (information pamphlets in treatment rooms), patient education and motivational support supplied through a digital CBTi coach, the digital CBTi coach was a peer support specialist working on the primary care mental health collaborative care team, the digital CBTi coach was trained by the research team, technical support and oversight of the digital CBTi coach by the research team. Additional members primary care mental health collaborative care team were educated by the research team to provide education to patients about digital CBTi. Multiple referral pathways to digital CBTi: consults to the digital CBTi Coach, warm handoffs to primary care mental health collaborative care team. Digital CBTi coach consults integrated Primary Care Workflow (Primary care provider placed consult in the medical record).
Period: Overall Study
Arm/Group | Phase 1: Implementation As Usual (Implementation Through Research Team) | Phase 2: Primary Care Coached Digital CBTi Implementation (Implementation Through Primary Care) | Phase 3: Primary Care Mental Health Collaborative Care Implementation
Started | 27 | 20 | 30
Completed | 25 | 19 | 26
Not Completed | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Implementation As Usual (Implementation Through Research Team) | Phase 2: Primary Care Coached Digital CBTi Implementation (Implementation Through Primary Care) | Phase 3: Primary Care Mental Health Collaborative Care Implementation | Total
Number analyzed (Participants) | 27 | 20 | 30 | 77
Age, Customized [Count of Participants; unit: Participants]
  <=55 | 8 | 7 | 7 | 22
  >55,<=65 | 9 | 4 | 9 | 22
  >65 | 10 | 9 | 14 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 6 | 11
  Male | 23 | 19 | 24 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/non-Hispanic | 21 | 13 | 24 | 58
  African American/Non-Hispanic | 2 | 4 | 3 | 9
  Hispanic | 3 | 2 | 2 | 7
  Other | 1 | 1 | 1 | 3
Any Mental Health Diagnosis [Count of Participants; unit: Participants]
  Any Mental Health Diagnosis | 12 | 8 | 15 | 35
  No Mental Health Diagnosis | 15 | 12 | 15 | 42
Number of Medical Diagnoses [Count of Participants; unit: Participants]
  <5 | 4 | 6 | 7 | 17
  >=5, <10 | 10 | 4 | 7 | 21
  >=10 | 13 | 10 | 16 | 39
Any Sedative-Hypnotic Prescription [Count of Participants; unit: Participants]
  Any Sedative-Hypnotic Prescription | 6 | 4 | 12 | 22
  No Sedative-Hypnotic Prescription | 21 | 16 | 18 | 55

OUTCOME MEASURES:

1. Primary Outcome: Program Engagement: Completion of the First Program Module
Description: The proportion of participants engaging in the program (completing at least one module) among the unique Veterans treated in VA Connecticut primary care over the respective intervention periods.
Time Frame: 3 weeks following subject enrollment
Population: Unique Veterans treated in VA Connecticut primary care over the respective intervention periods.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Implementation As Usual (Implementation Through Research Team): SHUTi digital CBTi Program was implemented in VACT primary care using implementation activities executed by the research team between June 2017 and January 2018 (8-months). Implementation activities included: Provider Education by the research team, Provider Reminders (information pamphlets in treatment rooms), Patient Advertising/Information (information pamphlets in treatment rooms), Single Referral Pathway Not Integrated Primary Care Workflow (Primary care provider contact research team for patient referral over email).
- Phase 2: Primary Care Coached Digital CBTi Implementation (Implementation Through Primary Care): SHUTi digital CBTi Program implemented in VACT primary care using implementation activities executed by primary care teams June 2018 and January 2019 (8-months). Implementation activities included: Provider Education by the research team, Provider Reminders (information pamphlets in treatment rooms), Patient Advertising/Information (information pamphlets in treatment rooms), patient education and motivational support supplied through a digital CBTi coach, the digital CBTi coach was a primary care nurse trained by the research team, technical support and oversight of the digital CBTi coach by the research team. Single Referral Pathway Not Integrated Primary Care Workflow.
- Phase 3: Primary Care Mental Health Collaborative Care Implementation: SHUTi digital CBTi Program implemented in VACT primary care using implementation activities executed by primary care teams April 2019 and November 2019 (8-months). Implementation activities included: Provider Education by the research team, Provider Reminders, Patient Advertising/Information, patient education and motivational support supplied through a digital CBTi coach, the digital CBTi coach was a peer support specialist working on the primary care mental health collaborative care team, the digital CBTi coach was trained by the research team, technical support and oversight of the digital CBTi coach by the research team. Additional members primary care mental health collaborative care team were educated to provide education about digital CBTi. Multiple referral pathways to digital CBTi: consults to the digital CBTi Coach, warm handoffs to primary care mental health collaborative care team. Digital CBTi coach consults integrated Primary Care Workflow.
Arm/Group | Phase 1: Implementation As Usual (Implementation Through Research Team) | Phase 2: Primary Care Coached Digital CBTi Implementation (Implementation Through Primary Care) | Phase 3: Primary Care Mental Health Collaborative Care Implementation
Number analyzed (Participants) | 12658 | 13592 | 13572
Participants | 17 | 12 | 16

2. Secondary Outcome: Program Completion
Description: Completion of all six modules of the program. The proportion of individuals completing all six modules among all individuals enrolled.
Time Frame: 10 Weeks following subject enrollment
Population: Individuals enrolled in the trial over the respective active implementation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Implementation As Usual (Implementation Through Research Team) | Phase 2: Primary Care Coached Digital CBTi Implementation (Implementation Through Primary Care) | Phase 3: Primary Care Mental Health Collaborative Care Implementation
Number analyzed (Participants) | 27 | 20 | 30
Participants | 10 | 7 | 7

3. Secondary Outcome: Provider Adoption
Description: The number of providers who made a referral to the SHUTi Program among the number of providers with the ability to make a referral.
Time Frame: Over each 8-month active implementation Phase
Population: Denominator of providers with the potential to make referrals over each period is estimated due to frequent provider transitions, changes to the referral process, and training programs within primary care.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Implementation As Usual (Implementation Through Research Team) | Phase 2: Primary Care Coached Digital CBTi Implementation (Implementation Through Primary Care) | Phase 3: Primary Care Mental Health Collaborative Care Implementation
Number analyzed (Participants) | 60 | 60 | 60
Participants | 31 | 26 | 34

4. Secondary Outcome: Insomnia Severity Index
Description: The ISI will be the primary clinical outcome and is a self-report seven-item measure that targets the subjective symptoms and functional consequences of insomnia. The outcome reported is the change in total ISI score from baseline to follow-up. All enrollees are analyzed as a single group regardless of implementation period. The Insomnia Severity Index to total is the sum on 7 questions scored 0 to 4 (minimum=0, Maximum=28). Higher scores indicate more severe insomnia.
Time Frame: At enrollment and 10 weeks following enrollment.
Population: All enrollees in the trial.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Enrollees: All enrollees are analyzed as a single group regardless of implementation period. The ISI will be the primary clinical outcome and is a self-report seven-item measure that targets the subjective symptoms and functional consequences of insomnia.
Arm/Group | All Enrollees
Number analyzed (Participants) | 70
score on a scale | 4.3 (5.6)

5. Other Pre Specified Outcome: Beck Depression Inventory
Description: The BDI is a secondary clinical outcome and is a self-report measure of depression severity. The outcome reported is the change in total BDI score from baseline to follow-up. All enrollees are analyzed as a single group regardless of implementation period. The BDI is a 21-item, self-report rating inventory of depression symptoms. Items receive a rating of zero to three and are summed linearly to create a score which ranges from 0 to 63. Higher score indicate more intense symptoms of depression.
Time Frame: At enrollment and 10 weeks following enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Enrollees: All enrollees are analyzed as a single group regardless of implementation period.
Arm/Group | All Enrollees
Number analyzed (Participants) | 70
score on a scale | 3.1 (5.5)

6. Other Pre Specified Outcome: Sedative-Hypnotic Medication Use
Description: The use of sedative-hypnotics will be measured by self-report of the type and dose of specific medications used in the last week. The outcome reported is the change in the reported total weekly number of sedative-hypnotic doses reported from baseline compared to follow-up.
Time Frame: At enrollment and 10 weeks following enrollment
Measure: Mean (Standard Deviation); unit: weekly sedative-hypnotic doses
Arm/Group | All Enrollees
Number analyzed (Participants) | 70
weekly sedative-hypnotic doses | 2.2 (6.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entire trial period between June 2017 and January 2020. This timeframe included the 3 periods of active implementation (when referrals could be made to the program) in addition to periods where subjects who had enrolled could actively engage in the SHUTi (up to 10 weeks after enrollment).
Description: Enrollment in this trial and engagement in the SHUTi program was determined to pose no greater that minimal risks to subjects. An adverse event was defined as an unfavorable medical occurrence that could be considered related to the participant's participation in the research.
Arm/Group | All Enrollees
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 0/77

LIMITATIONS AND CAVEATS:
The research team realized that implementation in phase 2 was not resulting in improved implementation outcomes over phase 1. Formative evaluation of implementation took place, and and additional implementation phase (phase 3) was added.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT03151083/Prot_SAP_000.pdf